CLINICAL TRIAL: NCT06647862
Title: A Randomized, Controlled, Double-Blind, Multicenter, Phase Ⅲ Study to Evaluate the Efficacy and Safety of IMM01 (Timdarpacept) in Combination With Azacitidine in Patients With Newly Diagnosed Chronic Myelomonocytic Leukemia (CMML1-2)
Brief Title: IMM01+Azacitidine VS Placebo +Azacitidine in Patients With Newly Diagnosed Chronic Myelomonocytic Leukemia (CMML1-2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMM01-010
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMM01 in combination with azacitidine (Experimental): One treatment cycle consists of 4 weeks (28 days). IMM01(timdarpacept) will be administered once weekly, and azacitidine will be administered from Day 1 to Day 7 of each cycle.
  Interventions: Drug: IMM01; Drug: Azacitidine
- placebo in combination with azacitidine (Placebo Comparator): One treatment cycle consists of 4 weeks (28 days). Placebo will be administered once weekly, and azacitidine will be administered on days 1-7 of each cycle.
  Interventions: Drug: Azacitidine; Drug: Placebo

INTERVENTIONS:
Drug: IMM01 — IV infusion
  Other Names: Timdarpacept
  Arms: IMM01 in combination with azacitidine
Drug: Azacitidine — subcutaneous injection
Drug: Placebo — IV infusion
  Arms: placebo in combination with azacitidine

SUMMARY:
This study is a randomized, controlled, double-blind, multicenter, phase Ⅲ clinical study to evaluate the efficacy of IMM01(timdarpacept) in combination with azacitidine versus placebo in combination with azacitidine in patients with newly diagnosed chronic leukemia monocytic (CMML1-2).Primary endpoint are Complete remission rate and Overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, regardless of gender;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
* Life expectancy ≥ 12 weeks;
* Patients with CMML diagnosed according to WHO 2016 criteria, including CMML-1 and CMML-2;
* White blood cell count ≤ 13×10⁹/L before the first treatment with the study drug (hydroxyurea and leukapheresis are allowed).
* Patients must be treatment-naïve to any systemic agents for CMML (e.g., azacitidine, decitabine,chemotherapy<1 cycle, and the washout period should be more than 28 days, which is acceptable.), allogeneic stem cell transplant for CMML. Note: During screening and study participation, subjects may continue oral corticosteroids for diseases other than CMML (e.g. asthma) at a stable daily dose equivalent to ≤ 10 mg prednisone. In addition, supportive care in the form of blood transfusions or growth factors is not considered prior therapy in this case and is permitted prior to and as needed during the study.

Exclusion Criteria:

* Previous treatment with anti-CD47 monoclonal antibody/SIRPα fusion protein;
* History of allogeneic stem cell transplant and other organ transplants; Patients who have undergone autologous haematopoietic stem cell transplant;
* Prior diagnosis of: therapy-related Myelodysplastic syndrome / Myeloproliferative neoplasm(MDS/MPN); MDS evolved from a pre-existing Myelodysplastic syndrome / Myeloproliferative neoplasm (MDS/MPN) ;other MDS/MPN including atypical chronic myeloid leukemia (aCML), juvenile myelomonocytic leukemia (JMML) and unclassifiable MDS/MPN. Patients positive for BCR-ABL fusion genes, PDGFRA, PDGFRB, and FGFR1 rearrangements need to be excluded;
* Current or history of central nervous system (CNS) leukemia, extramedullary leukemia(excluding: Enlarged spleen, enlarged liver, enlarged lymph nodes), or myeloid sarcoma;
* Diagnosis of other malignant neoplasms within 3 years prior to the first dose. Exceptions: a. Radically treated cervical carcinoma in situ or non-melanoma skin cancer,Surgery-cured prostate cancer and papillary thyroid cancer; b. a second primary cancer that has been curatively treated and has no recurrence within three years;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2029-10-24 (Estimated)

PRIMARY OUTCOMES:
Complete remission( CR) rate | approximately 24 months
  CR rate: CR rate determined by Independent Review Committee (IRC) based on IWG2006 MDS efficacy evaluation criteria;
Overall survival (OS) | approximately 24 months
  Overall survival (OS): Time from randomization to death from any cause;

SECONDARY OUTCOMES:
Event-free survival(EFS) | approximately 24 months
  Time from randomization to transformation to AML or death from any cause, whichever occurs first
Progression-free survival(PFS) | approximately 24 months
  Time from randomization to transformation to AML or death from any cause, whichever occurs first
Time to response (TTR) | approximately 24 months
  time from first dose to first occurrence of CR, partial remission (PR), marrow complete remission (mCR) ± hematologic improvement (HI), HI, assessed by IRC and investigators, respectively
overall response rate(ORR) | approximately 24 months
  is defined as the proportion of the analysis population achieving CR, PR, mCR±HI, or HI
Duration of response(DOR) | approximately 24 months
  is defined as the time from the first occurrence of CR, PR, mCR±HI, or HI to disease progression or death from any cause, whichever occurs first
Red blood cell transfusion independence (RTI) | approximately 24 months
  the proportion of patients who did not receive red blood cell (or whole blood) transfusion for 8 consecutive weeks during the study treatment period among patients who required transfusion at baseline.
Complete remission(CR) rate | approximately 24 months
  CR rate determined by IRC based on IWG2006 MDS efficacy evaluation criteria assessed by the investigator;
Time to transformation to acute myeloid leukemia | approximately 24 months
  Time from initiation of study treatment to transformation to AML; defined as ≥ 20% blasts in the bone marrow or peripheral blood by manual differential count, according to the 2016 WHO classification criteria.

CONTACTS AND LOCATIONS:
Overall Officials: zhijian xiao, PHD, Principal Investigator — Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College; Hongyan Tong, PHD, Principal Investigator — Zhejiang University
Locations (43):
- China (43):
  - Anhui Provincial Hospital, Hefei, Anhui
  - China-Japan Friendship Hospita, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - First Hospital of Lanzhou University, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Gaungxi
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Zhujiang Hospital of Southern Medical University, Zhujiang, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangzhou
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Hebei University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin First Hospital, Harbin, Heilongjiang
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Zhengzhou, Henan
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital Affiliated to Wuhan University, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Changzhou First People's Hospital, Changzhou, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Zhongda Hospital affiliated to Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiangsu Subei People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shaanxi Provincial People's Hospital, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College;, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Peking University People's Hospital, Beijing
  - Tianjin People's Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No